CLINICAL TRIAL: NCT06615739
Title: PMCF Study to Provide Safety, Performance and Clinical Benefits Data of the Comprehensive Segmental Revision System (SRS) Regenerex Tissue Attachment Augments - A Retrospective Enrollment and Prospective Follow-up Consecutive Series Study
Brief Title: Comprehensive SRS Regenerex Tissue Attachment
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2024-12E
Record Dates: First submitted 2024-09-18; First posted 2024-09-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Arthroplasty Complications; Osteo Arthritis Shoulders
Keywords: Medical Device; Safety; Performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Comprehensive Regenerex Tissue Attachment Augments: Regenerex Tissue Attachment Augments were used in combination with the Comprehensive Segmental Revision system
  Interventions: Device: Regenerex Tissue Attachment Augments

INTERVENTIONS:
Device: Regenerex Tissue Attachment Augments — Patient will have been previously implanted with Regenerex Tissue Attachment Augments in combination with the Comprehensive Segmental Revision System

SUMMARY:
The objective of this retrospective and prospective consecutive series data collection is to confirm safety, performance, and clinical benefits of the Comprehensive SRS Regenerex Tissue Attachment Augments when used for limb salvage arthroplasty.

DETAILED DESCRIPTION:
Consecutive subjects implanted with Comprehensive SRS Regenerex Tissue Attachment Augments according to the approved indications, with the longest-term follow-up possible, will be identified and invited to participate in the study.

The primary objective is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications, and adverse events. Relation of the events to the implant and/or procedure should be specified.

The study will include one site. There will be a maximum of 103 patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient must be willing and able to follow directions.
* The Comprehensive Segmental Revision System was used in cases of:

  1. Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
  2. Revision where other devices or treatments have failed.
  3. Correction of functional deformity.
  4. Oncology applications including bone loss due to tumor resection.
* Proximal or total humeral replacement, for: Treatment of acute or chronic fractures with humeral head (shoulder) involvement, which are unmanageable using other treatment methods.
* Distal or total humeral replacement for: Treatment of acute or chronic fractures with humeral epicondyle (elbow) involvement, which are unmanageable using other treatment methods.
* Biomet Comprehensive Segmental Revision System was used in a reverse application in patients whose shoulder joint has a grossly deficient rotator cuff with severe arthropathy and/or previously failed shoulder joint replacement with a grossly deficient rotator cuff for proximal humeral replacement. The patient must be anatomically and structurally suited to receive the implants and a functional deltoid muscle is necessary.
* The Comprehensive Segmental Revision System was used with bone cement in distal humeral and total humeral applications.
* Regenerex Tissue Attachment Augments were used in combination with the Comprehensive Segmental Revision System

Exclusion Criteria:

* Absolute contraindications:

  * Infection
  * Sepsis
  * Osteomyelitis
  * Patient is a prisoner
  * Patient is a current alcohol or drug abuser
  * Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent
  * Patient is unwilling to consent
* Relative contraindications:

  * Uncooperative patient or patient with neurologic disorders who is incapable of following directions
  * Osteoporosis
  * Metabolic disorders which may impair bone formation
  * Osteomalacia
  * Distant foci of infections which may spread to the implant site
  * Vascular insufficiency, muscular atrophy, or neuromuscular disease
* The Comprehensive Segmental Revision System was used in a reverse shoulder application in patients receiving radiation therapy
* The Comprehensive Segmental Revision System was used without bone cement in distal humeral and total humeral applications.
* Regenerex Tissue Attachment Augments weren't used during the patient's surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must meet the inclusion criteria to be enrolled into the study. Subjects who meet any of the exclusion criteria should not be enrolled into the study.
  The study population will comprise a consecutive cohort of up to 103 subjects implanted using the Comprehensive SRS Regenerex Tissue Attachment Augments.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Kaplan Meier Implant Survivorship | Up to 10 Years
  This will be established by recording the incidence and frequency of device revisions. Kaplan-Meier survival analysis is a statistical method that estimates survival rates over time and accounts for factors that can affect implant survival.
Safety Assessement | Up to 10 Years
  This will be established by recording the incidence and frequency of complications and adverse events. Relation of the events to the implant and/or procedure will be specified.

SECONDARY OUTCOMES:
Assessment of performance and clinical benefits by recording patient reported QuickDASH | Up to 10 Years
  QuickDASH, or Quick Disabilities of the Arm, Shoulder, and Hand, is a questionnaire that measures the impact of upper limb musculoskeletal disorders on physical function and symptoms.
  The QuickDASH has 11 items that cover six domains:
  Daily activities: How much difficulty the patient has performing physical activities Symptoms: How severe the patient's pain and tingling is Social function: How the patient's problem affects their social activities Work function: How the patient's problem affects their work Sleep: How the patient's problem affects their sleep Confidence: How the patient's problem affects their confidence
  Each item is rated on a 5-point Likert scale, with 1 being no difficulty and 5 being unable. The score is then converted to a 100-point scale, with 100 representing the greatest disability.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (1):
- Toman Orthopedics and Sports Med, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shared due to this being a single center retrospective enrollment/prospective FUP with one single reference point. Additionally, data is being collected for EU regulatory purposes.